CLINICAL TRIAL: NCT02631369
Title: Measuring Cyclotorsion on Scanning Laser Ophthalmoscopy (SLO)-Fundus Photographs Using the Integrated Algorithm by Heidelberg Spectralis
Brief Title: Measuring Cyclotorsion on Scanning Laser Ophthalmoscopy (SLO)-Fundus Photographs
Acronym: CySLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KEK-ZH-Nr. 2014-0404
Record Dates: First submitted 2015-12-09; First posted 2015-12-16 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Trochlear Nerve Diseases
MeSH Terms: conditions — Trochlear Nerve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- inter- & intrarater reliability study (Experimental): pre-study: inter- and intrarater reliability study in 30 healthy subjects, interventions: SLO-fundus photographs using the integrated algorithm by Heidelberg Spectralis OCT (optical coherence tomography) device
  Interventions: Device: Heidelberg Spectralis OCT device
- cyclotorsion in forth nerve palsy (Experimental): measurement of cyclotorsion on SLO-fundusphoto in 20 patients forth nerve palsy interventions: SLO-fundus photographs using the integrated algorithm by Heidelberg Spectralis OCT (optical coherence tomography) device
  Interventions: Device: Heidelberg Spectralis OCT device
- cyclotorsion in healthy subjects (Experimental): measurement of cyclotorsion on SLO-fundusphoto in 30 healthy subjects to be compared to patients with forth nerve palsy interventions: SLO-fundus photographs using the integrated algorithm by Heidelberg Spectralis OCT (optical coherence tomography) device
  Interventions: Device: Heidelberg Spectralis OCT device

INTERVENTIONS:
Device: Heidelberg Spectralis OCT device

SUMMARY:
Pre-Study: Evaluation of the inter- and intrarater reliability of the integrated algorithm by Heidelberg Spectralis for measuring cyclotorsion on SLO-fundus fotographs, and assessment of the influence of measuring with or without eye tracker.

Study: Comparison of cyclotorsion measurements in patients with forth nerve palsy and in healthy controls on SLO-fundus fotographs using the integrated algorithm by Heidelberg Spectralis

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* best corrected visual acuity ≥ 0.8

Exclusion Criteria:

* strabismus except for forth nerve palsy
* previous strabismus surgery
* monocle
* best corrected visual acuity ≤ 0.6
* hyperopia or myopia > 6dpt

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
pre-study: reliability of repeated measurements of excyclotorsion in degrees on SLO-fundus fotographs | 3 months
  pre-study: inter- and intrarater reliability of the device with or without eye tracker; excyclotorsion in degrees (based on the line crossing the fovea and the center of the optic nerve head) as provided by the integrated algorithm by Heidelberg Spectralis
study: excyclotorsion in degrees on SLO-fundus fotographs | 12 months
  study: comparison of cyclotorsion measurements in healthy controls compared to patients with forth nerve palsy; excyclotorsion in degrees (based on the line crossing the fovea and the center of the optic nerve head) as provided by the integrated algorithm by Heidelberg Spectralis

SECONDARY OUTCOMES:
study: excyclotorsion in degrees on tangent screen, double maddox and fundus photographs | 12 months
  validation of the cyclotorsion measurement with the Heidelberg Spectralis device against tangent screen [degrees], double maddox [degrees] and fundus photographs [degrees]

CONTACTS AND LOCATIONS:
Overall Officials: Ghislaine L Traber, MD, Principal Investigator — University Hospital Zurich, Dept of Ophthalmology
Locations (1):
- University Hospital Zurich, Dept of Ophthalmology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Lengwiler F, Rappoport D, Jaggi GP, Landau K, Traber GL. Reliability of Cyclotorsion measurements using Scanning Laser Ophthalmoscopy imaging in healthy subjects: the CySLO study. Br J Ophthalmol. 2018 Apr;102(4):535-538. doi: 10.1136/bjophthalmol-2017-310396. Epub 2017 Aug 1. PMID 28765146